CLINICAL TRIAL: NCT03215472
Title: DASH Cloud: Using Digital Health to Improve Adherence to the DASH Diet Among Women at Risk for Cardiovascular Disease
Brief Title: DASH Cloud: Using Digital Health to Improve Adherence to the DASH Diet Among Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081972
Record Dates: First submitted 2017-06-20; First posted 2017-07-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2018-03

CONDITIONS: Diet Modification; Hypertension; Women's Health; Cardiovascular Diseases; Digital Health
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 3-month randomized controlled trial to test the initial feasibility of DASH Cloud, a digital health intervention for women at risk for CVD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH Cloud intervention (Experimental): In group 1, participants will be instructed to input their dietary intake daily for three months using the Nutritionix app. A participant's data will automatically be uploaded from the Nutritionix app via the API that links the device with DASH Cloud. DASH Cloud will run an algorithm and send daily or weekly feedback text messages reflecting DASH adherence. The intervention components include tailored feedback texts, and behavioral skills training videos.
  Interventions: Other: DASH Cloud
- Dash Light (Experimental): Group 2 participants will be asked to use the Nutritionix app daily and receive publicly available written materials on the DASH diet.
  Interventions: Other: Nutritionix Track app

INTERVENTIONS:
Other: DASH Cloud — With DASH Cloud, the investigators will ask participants to track their diet daily using a commercial diet tracking app. The investigators will retrieve the diet data on our DASH Cloud platform and provide tailored feedback about a participant's DASH adherence via fully automated daily or weekly text messages. These feedback messages will describe both an individual's absolute performance and change over time. The investigators also include theory-driven tailored content that reinforces successes, offers motivational strategies, and offers short behavior change tips.
  Arms: DASH Cloud intervention
Other: Nutritionix Track app — DASH Light Control participants will be asked to use the Nutritionix app daily and receive publicly available written materials on the DASH diet.
  Other Names: DASH Light
  Arms: Dash Light

SUMMARY:
This study will test whether a digital health intervention (DASH Cloud) using smartphones can improve diet quality among women at risk for cardiovascular disease. The DASH (Dietary Approaches to Stop Hypertension) Diet has been proven to lower blood pressure, yet dissemination efforts remain poor. This study aims to use technology to improve adherence to DASH.

DETAILED DESCRIPTION:
Specifically, this study aims to

1. To test the feasibility of the DASH Cloud intervention compared to education control among women with prehypertension and hypertension via a 3-month randomized controlled trial.
2. To evaluate the preliminary efficacy of the DASH Cloud intervention relative to education control on blood pressure, weight and medication adherence at 3 months.

This study will enroll 50 adult women aged 21-70 with pre-hypertension or hypertension in a 3-month randomized controlled trial to test the initial feasibility of DASH Cloud. Women will be randomized to either the DASH Cloud intervention or DASH Light and followed up 3 months post randomization. The investigators will recruit participants from the Durham, NC area.

Women randomized to the DASH Cloud intervention will be asked to track their diet daily using a smartphone diet tracking app. Based on the foods/beverages entered, the intervention will send daily or weekly text messages with feedback about DASH adherence and information videos about how to follow DASH. Women randomized to DASH Light will also be asked to track their diet using the smartphone diet tracking app and will receive basic informational materials about DASH.

ELIGIBILITY:
Inclusion Criteria:

* ages 21-70 years; BMI >18.5 kg/m2
* on antihypertensive medication or systolic blood pressure 120-159 mmHg and/or diastolic blood pressure of 80-99
* current use of a smartphone and willingness to be texted daily or weekly
* an email account; spoken and written English fluency.

Exclusion Criteria:

* CVD event in prior 6 months
* active malignancy; active psychosis or recent psychiatric institutionalization
* current pregnancy or lactation
* current participation in a similar trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Adherence to the DASH Diet | 3 months
  Dietary intake data will be collected using NCI's Automated Self-Administered 24-hour Recall tool.

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline, 3 months
  Blood pressure will be measured at baseline and 3 months in the upper arm in triplicate at 1-minute intervals. Measurements will be obtained using the validated Omron HEM-907XL blood pressure monitor.
Change in Weight | Baseline, 3 months
  Weight will be collected in kilograms at baseline and 3 months using a calibrated digital scale.
Engagement | 3 months
  Utilization of intervention component (daily diet tracking using Nutritionix app) at 3 months. This will be measured by the proportion of participants completing daily dietary self-monitoring.
Engagement | 3 months
  Utilization of intervention component (review of skills training videos) at 3 months. This will be measured by the number of clicks to skills training via video tracking software.

CONTACTS AND LOCATIONS:
Overall Officials: Dori M Steinberg, PhD, RD, Principal Investigator — Duke University
Locations (1):
- The Sarah W. Stedman Nutrition and Metabolism Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kay MC, Miller HN, Askew S, Spaulding EM, Chisholm M, Christy J, Yang Q, Steinberg DM. Patterns of Engagement With an Application-Based Dietary Self-Monitoring Tool Within a Randomized Controlled Feasibility Trial. AJPM Focus. 2022 Sep 29;1(2):100037. doi: 10.1016/j.focus.2022.100037. eCollection 2022 Dec. PMID 37791242
- [Derived] Steinberg DM, Kay MC, Svetkey LP, Askew S, Christy J, Burroughs J, Ahmed H, Bennett GG. Feasibility of a Digital Health Intervention to Improve Diet Quality Among Women With High Blood Pressure: Randomized Controlled Feasibility Trial. JMIR Mhealth Uhealth. 2020 Dec 7;8(12):e17536. doi: 10.2196/17536. PMID 33284116

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03215472/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03215472/SAP_001.pdf